CLINICAL TRIAL: NCT05837000
Title: Role of Adding Dexmedetomidine, Ketamine and Magnesium Sulphate to Caudal Block as Preemptive Analgesia in Hypospadias Repair in Pediatrics: a Randomized Double-blinded Trial
Brief Title: Dexmedetomidine, Ketamine and Magnesium Sulphate in Caudal Block for Hypospadias Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Gamal Hendawy Shams, Lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 51- 2 - 16
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Preemptive Analgesia; Dexmedetomidine; Ketamine; Magnesium Sulphate; Hypospadias; Pediatrics
MeSH Terms: conditions — Hypospadias | interventions — Dexmedetomidine; Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): 0.5 ml/kg bupivacaine 0.25% + 1μg/kg dexmedetomidine caudally
  Interventions: Drug: Dexmedetomidine
- Ketamine (Experimental): 0.5 ml/kg bupivacaine 0.25% + 1μg/kg dexmedetomidine caudally
  Interventions: Drug: Ketamine
- Magnesium sulphate (Experimental): 0.5ml/kg bupivacaine 0.25% + 1ml volume containing 50mg of magnesium caudally.
  Interventions: Drug: Magnesium sulphate

INTERVENTIONS:
Drug: Dexmedetomidine — Patient will receive 0.5 ml/kg bupivacaine 0.25% + 1μg/kg dexmedetomidine caudally
  Arms: Dexmedetomidine
Drug: Ketamine — Patient will receive 0.5ml/kg bupivacaine 0.25% + 0.5mg/kg ketamine caudally
  Arms: Ketamine
Drug: Magnesium sulphate — Patient will receive 0.5ml/kg bupivacaine 0.25% + 1ml volume containing 50mg of magnesium caudally.
  Arms: Magnesium sulphate

SUMMARY:
Caudal epidural block is a rapid, reliable, and safe technique that can be used with general anesthesia for intraoperative and postoperative analgesia in pediatric patients Ketamine is a selective antagonist of N-methyl-D-aspartate (NMDA) receptor, an ionotropic glutamate receptor.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-7 years
* American Society of Anesthesiologists (ASA) classification I and II, undergoing hypospadias repair.

Exclusion Criteria:

* Developmental delay
* Psychological or neurological disorders
* Difficult airway
* Hyperactive airway disease or children in whom caudal block was contraindicated (e.g., infection at the site of block, bleeding disorder, or abnormalities of the sacrum).

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — males
Enrollment: 75 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
First time of rescue analgesia requirement | 24 hours postoperatively
  If the FLACC score is ≥ 4, pethidine 1 mg/kg. The first time to require analgesia will be calculated (the time from caudal block to the first time to pethidine injection).

SECONDARY OUTCOMES:
Total consumption of rescue analgesia | 24 hours postoperatively
  If the FLACC score is ≥ 4, pethidine 1 mg/kg. The total pethidine consumption of patients require analgesia in the first 24 h postoperative will be calculated.
Pain score | 24 hours postoperatively
  FLACC scale will used for postoperative pain assessment. This scale ranges from 0 to 10 where 0 represents no pain and 10 represents worst possible pain
The incidence of adverse effects | 24 hours postoperatively
  Hypotension bradycardia, respiratory depression and vomiting will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kafrelsheikh University, Principal Investigator — Research ethics committee - Kafrelsheikh University
Locations (1):
- Karelsheikh University Hospital, Kafr ash Shaykh, Karelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon Reasonable request from the corresponding author for one year after study completion
Supporting Information: Study Protocol
Time Frame: The data will be available for one year after study completion
Access Criteria: The data will be available upon Reasonable request from the corresponding author.

REFERENCES:
- Available data/document: Study Protocol: MKSU 51- 2 _ 16 — http://kfs.edu.eg/engkfs/